CLINICAL TRIAL: NCT05786222
Title: Permanent Supportive Housing Overdose Prevention (POP) Study: A Hybrid Type 3 Stepped Wedge Randomized Controlled Trial
Brief Title: Permanent Supportive Housing Overdose Prevention
Acronym: POP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-00098
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Overdose
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cluster 1 (Experimental): Buildings randomized to Cluster 1 will receive the CSH-delivered intervention at Months 2-7. Tenant surveys will be administered 1 month prior to and 12 months following the start of the intervention period.
  At all clusters, an all-staff survey will be administered at Months 1, 8, 15, 22, and 29. A sustainment survey will be administered to selected staff-leaders in the 8th month following the end of the intervention period.
  Interventions: Behavioral: CSH-Delivered Overdose Prevention Support
- Cluster 2 (Experimental): Buildings randomized to Cluster 2 will receive the CSH-delivered intervention at Months 9-14. Tenant surveys will be administered 1 month prior to and 12 months following the start of the intervention period.
  At all clusters, an all-staff survey will be administered at Months 1, 8, 15, 22, and 29. A sustainment survey will be administered to selected staff-leaders in the 8th month following the end of the intervention period.
  Interventions: Behavioral: CSH-Delivered Overdose Prevention Support
- Cluster 3 (Experimental): Buildings randomized to Cluster 3 will receive the CSH-delivered intervention at Months 16-21. Tenant surveys will be administered 1 month prior to and 12 months following the start of the intervention period.
  At all clusters, an all-staff survey will be administered at Months 1, 8, 15, 22, and 29. A sustainment survey will be administered to selected staff-leaders in the 8th month following the end of the intervention period.
  Interventions: Behavioral: CSH-Delivered Overdose Prevention Support
- Cluster 4 (Experimental): Buildings randomized to Cluster 3 will receive the CSH-delivered intervention at Months 23-28. Tenant surveys will be administered 1 month prior to and 12 months following the start of the intervention period.
  At all clusters, an all-staff survey will be administered at Months 1, 8, 15, 22, and 29. A sustainment survey will be administered to selected staff-leaders in the 8th month following the end of the intervention period.
  Interventions: Behavioral: CSH-Delivered Overdose Prevention Support

INTERVENTIONS:
Behavioral: CSH-Delivered Overdose Prevention Support — Corporation for Supportive Housing (CSH) will deliver technical support for overdose (OD) prevention in the participating PSH buildings using a package of core implementation strategies: PSH Overdose Prevention (POP) Toolkit (an implementation manual/blueprint for overdose prevention practices); Implementation Champions (staff and tenants in each PSH building will be selected as implementation champions who support implementation and sustainment of OD prevention practices in their buildings); practice facilitation (the practice facilitator [a trained CSH employee] will work with the tenant and staff champions in small group workshops and coaching sessions, building their capacity and supporting their work toward implementation of building OD prevention practices); learning collaboratives (PSH buildings starting the intervention at the same time will attend learning collaborative meetings).

SUMMARY:
Permanent supportive housing (PSH), the gold standard intervention for ending chronic homelessness, has expanded rapidly across the U.S. in recent years. Due to a confluence of individual and environmental risk factors, PSH tenants face heightened risk for overdose. While evidence-based practices to prevent overdose exist, they have not been broadly implemented in PSH settings. This study will address this research to practice gap by studying the implementation of evidence-based practices to prevent overdose in 20 PSH buildings in New York. In a community-partnered stepped wedge randomized controlled trial, the investigators will study a package of implementation strategies that includes an implementation toolkit, tenant and staff implementation champions, limited practice facilitation, and learning collaboratives. Outcomes will be examined using surveys and qualitative interviews with PSH tenants and staff; observation; and analysis of Medicaid claims data.

DETAILED DESCRIPTION:
This single-center study is a hybrid type 3 trial with a stepped wedge cluster randomized controlled trial design, with primary objectives of studying implementation of overdose prevention practices in PSH and secondary objectives of examining effectiveness on clinically relevant outcomes and multilevel factors influencing implementation. Twenty participating PSH building sites will be randomized into four intervention clusters of five buildings each. With the stepped wedge design, all clusters of study PSH buildings will begin in the control condition. Clusters are randomly assigned to receive the intervention at different times, with all eventually receiving the six-month implementation strategy package intervention from Corporation for Supportive Housing (CSH). Study investigators will survey PSH building tenants and staff; conduct observation of building policies and procedures; analyze tenant Medicaid data; and interview staff and tenants.

ELIGIBILITY:
Inclusion Criteria:

Tenant surveys: To be eligible to participate in the tenant survey part of this study, an individual must:

* Be a supportive housing tenant in a participating building
* Be at least 18 years old
* Be able to read and respond to a survey in English or Spanish

Staff surveys: To be eligible to participate in the staff survey part of this study, an individual must work for a participating PSH building (or have worked for one in the past 6 months). All PSH building staff are at least 18 years old and are able to read and respond to a survey in English. Staff surveys will begin with a question confirming eligibility.

Qualitative interviews: To be eligible to participate in the qualitative interview part of this study, an individual must:

* Work for or live in a participating PSH building
* Serve as staff (including leaders) or tenant implementation champion
* Be at least 18 years old
* Speak and understand English

Medicaid data analysis: Identifying information for all tenants in participating buildings (to be provided to the study team by buildings as described in a bilaterally signed information sharing agreement) will be used to conduct a match with Medicaid administrative data.

Exclusion Criteria:

Children under the age of 18 years old will be excluded, including from the Medicaid data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Fidelity Checklist Score | Month 1
  Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.
Fidelity Checklist Score | Month 8
  Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.
Fidelity Checklist Score | Month 15
  Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.
Fidelity Checklist Score | Month 22
  Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.
Fidelity Checklist Score | Month 29
  Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.

SECONDARY OUTCOMES:
Intervention Appropriateness Measure (IAM) Score | Month 1
  1-item assessment of intervention appropriateness (adapted from Weiner, et al.) for each of three overdose prevention categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Intervention Appropriateness Measure (IAM) Score | Month 8
  1-item assessment of intervention appropriateness (adapted from Weiner, et al.) for each of three overdose prevention categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Intervention Appropriateness Measure (IAM) Score | Month 15
  1-item assessment of intervention appropriateness (adapted from Weiner, et al.) for each of three overdose prevention categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Intervention Appropriateness Measure (IAM) Score | Month 22
  1-item assessment of intervention appropriateness (adapted from Weiner, et al.) for each of three overdose prevention categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Intervention Appropriateness Measure (IAM) Score | Month 29
  1-item assessment of intervention appropriateness (adapted from Weiner, et al.) for each of three overdose prevention categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Feasibility of Intervention Measure (FIM) Score | Month 1
  1-item assessment of intervention feasibility (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Feasibility of Intervention Measure (FIM) Score | Month 8
  1-item assessment of intervention feasibility (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Feasibility of Intervention Measure (FIM) Score | Month 15
  1-item assessment of intervention feasibility (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Feasibility of Intervention Measure (FIM) Score | Month 22
  1-item assessment of intervention feasibility (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Feasibility of Intervention Measure (FIM) Score | Month 29
  1-item assessment of intervention feasibility (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Brief Opioid Overdose Knowledge (BOOK) Survey Score | Month 1
  BOOK is a 12-item assessment of opioid overdose knowledge (Dunn, et al.) administered to staff. For each item, staff select either "True" or "False." The total score ranges from 0-12; higher scores indicate greater opioid overdose knowledge.
Brief Opioid Overdose Knowledge (BOOK) Survey Score | Month 8
  BOOK is a 12-item assessment of opioid overdose knowledge (Dunn, et al.) administered to staff. For each item, staff select either "True" or "False." The total score ranges from 0-12; higher scores indicate greater opioid overdose knowledge.
Brief Opioid Overdose Knowledge (BOOK) Survey Score | Month 15
  BOOK is a 12-item assessment of opioid overdose knowledge (Dunn, et al.) administered to staff. For each item, staff select either "True" or "False." The total score ranges from 0-12; higher scores indicate greater opioid overdose knowledge.
Brief Opioid Overdose Knowledge (BOOK) Survey Score | Month 22
  BOOK is a 12-item assessment of opioid overdose knowledge (Dunn, et al.) administered to staff. For each item, staff select either "True" or "False." The total score ranges from 0-12; higher scores indicate greater opioid overdose knowledge.
Brief Opioid Overdose Knowledge (BOOK) Survey Score | Month 29
  BOOK is a 12-item assessment of opioid overdose knowledge (Dunn, et al.) administered to staff. For each item, staff select either "True" or "False." The total score ranges from 0-12; higher scores indicate greater opioid overdose knowledge.
Perceived Stigma Toward Substance Users Scale Score | Month 1
  8-item assessment of perceived stigma toward substance users (Luoma, et al.). Survey is administered to staff. Each item is ranked on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The score is the sum of responses (with some items reverse-scored). The total score ranges from 8-32, with higher scores indicating greater perceived stigma.
Perceived Stigma Toward Substance Users Scale Score | Month 8
  8-item assessment of perceived stigma toward substance users (Luoma, et al.). Survey is administered to staff. Each item is ranked on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The score is the sum of responses (with some items reverse-scored). The total score ranges from 8-32, with higher scores indicating greater perceived stigma.
Perceived Stigma Toward Substance Users Scale Score | Month 15
  8-item assessment of perceived stigma toward substance users (Luoma, et al.). Survey is administered to staff. Each item is ranked on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The score is the sum of responses (with some items reverse-scored). The total score ranges from 8-32, with higher scores indicating greater perceived stigma.
Perceived Stigma Toward Substance Users Scale Score | Month 22
  8-item assessment of perceived stigma toward substance users (Luoma, et al.). Survey is administered to staff. Each item is ranked on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The score is the sum of responses (with some items reverse-scored). The total score ranges from 8-32, with higher scores indicating greater perceived stigma.
Perceived Stigma Toward Substance Users Scale Score | Month 29
  8-item assessment of perceived stigma toward substance users (Luoma, et al.). Survey is administered to staff. Each item is ranked on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The score is the sum of responses (with some items reverse-scored). The total score ranges from 8-32, with higher scores indicating greater perceived stigma.
Tenant Substance-Use-Related Emergency Department Visits | Month 1
  Data derived from NY Medicaid data.
Tenant Substance-Use-Related Emergency Department Visits | Month 8
  Data derived from NY Medicaid data.
Tenant Substance-Use-Related Emergency Department Visits | Month 15
  Data derived from NY Medicaid data.
Tenant Substance-Use-Related Emergency Department Visits | Month 22
  Data derived from NY Medicaid data.
Tenant Substance-Use-Related Emergency Department Visits | Month 29
  Data derived from NY Medicaid data.
Tenant Substance-Use-Related Emergency Department Visits | Month 35
  Data derived from NY Medicaid data.
Tenant Receipt of Medication for Opioid Use Disorder (MOUD) | Month 1
  Data derived from NY Medicaid data.
Tenant Receipt of Medication for Opioid Use Disorder (MOUD) | Month 8
  Data derived from NY Medicaid data.
Tenant Receipt of Medication for Opioid Use Disorder (MOUD) | Month 15
  Data derived from NY Medicaid data.
Tenant Receipt of Medication for Opioid Use Disorder (MOUD) | Month 22
  Data derived from NY Medicaid data.
Tenant Receipt of Medication for Opioid Use Disorder (MOUD) | Month 29
  Data derived from NY Medicaid data.
Tenant Receipt of Medication for Opioid Use Disorder (MOUD) | Month 35
  Data derived from NY Medicaid data.
Tenant Receipt of Specialty Substance Use Disorder (SUD) Treatment | Month 1
  Data derived from NY Medicaid data. Specialty SUD treatment includes outpatient, inpatient, and detoxification.
Tenant Receipt of Specialty Substance Use Disorder (SUD) Treatment | Month 8
  Data derived from NY Medicaid data. Specialty SUD treatment includes outpatient, inpatient, and detoxification.
Tenant Receipt of Specialty Substance Use Disorder (SUD) Treatment | Month 15
  Data derived from NY Medicaid data. Specialty SUD treatment includes outpatient, inpatient, and detoxification.
Tenant Receipt of Specialty Substance Use Disorder (SUD) Treatment | Month 22
  Data derived from NY Medicaid data. Specialty SUD treatment includes outpatient, inpatient, and detoxification.
Tenant Receipt of Specialty Substance Use Disorder (SUD) Treatment | Month 29
  Data derived from NY Medicaid data. Specialty SUD treatment includes outpatient, inpatient, and detoxification.
Tenant Receipt of Specialty Substance Use Disorder (SUD) Treatment | Month 35
  Data derived from NY Medicaid data. Specialty SUD treatment includes outpatient, inpatient, and detoxification.
Adoption Checklist Score | Month 1
  20-item checklist assessing building adoption of each overdose prevention practice. Checklist is included in a subset of staff surveys. Buildings will receive an adoption checklist score of 0 (not adopted) or 1 (adopted) for each of 20 overdose prevention practices. The total score is the sum of responses and ranges from 0-20, with higher scores indicating greater adoption.
Adoption Checklist Score | Month 8
  20-item checklist assessing building adoption of each overdose prevention practice. Checklist is included in a subset of staff surveys. Buildings will receive an adoption checklist score of 0 (not adopted) or 1 (adopted) for each of 20 overdose prevention practices. The total score is the sum of responses and ranges from 0-20, with higher scores indicating greater adoption.
Adoption Checklist Score | Month 15
  20-item checklist assessing building adoption of each overdose prevention practice. Checklist is included in a subset of staff surveys. Buildings will receive an adoption checklist score of 0 (not adopted) or 1 (adopted) for each of 20 overdose prevention practices. The total score is the sum of responses and ranges from 0-20, with higher scores indicating greater adoption.
Adoption Checklist Score | Month 22
  20-item checklist assessing building adoption of each overdose prevention practice. Checklist is included in a subset of staff surveys. Buildings will receive an adoption checklist score of 0 (not adopted) or 1 (adopted) for each of 20 overdose prevention practices. The total score is the sum of responses and ranges from 0-20, with higher scores indicating greater adoption.
Adoption Checklist Score | Month 29
  20-item checklist assessing building adoption of each overdose prevention practice. Checklist is included in a subset of staff surveys. Buildings will receive an adoption checklist score of 0 (not adopted) or 1 (adopted) for each of 20 overdose prevention practices. The total score is the sum of responses and ranges from 0-20, with higher scores indicating greater adoption.
Acceptability of Intervention Measure (AIM) Score | Month 1
  1-item assessment of intervention acceptability (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Acceptability of Intervention Measure (AIM) Score | Month 8
  1-item assessment of intervention acceptability (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Acceptability of Intervention Measure (AIM) Score | Month 15
  1-item assessment of intervention acceptability (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Acceptability of Intervention Measure (AIM) Score | Month 22
  1-item assessment of intervention acceptability (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Acceptability of Intervention Measure (AIM) Score | Month 29
  1-item assessment of intervention acceptability (adapted from Weiner, et al.) for each of the three overdose prevention practice categories, administered to staff and rated on a Likert scale from 1 (completely disagree) to 5 (completely agree).
Organizational Priority Measure Score | Month 1
  7-item assessment of organizational priority (adapted from Klein, et al.) administered to staff and rated on a Likert scale from 1 (not true) to 5 (definitely true). The total score is the sum of responses and ranges from 7 to 35; higher scores indicate higher organizational priority.
Organizational Priority Measure Score | Month 8
  7-item assessment of organizational priority (adapted from Klein, et al.) administered to staff and rated on a Likert scale from 1 (not true) to 5 (definitely true). The total score is the sum of responses and ranges from 7 to 35; higher scores indicate higher organizational priority.
Organizational Priority Measure Score | Month 15
  7-item assessment of organizational priority (adapted from Klein, et al.) administered to staff and rated on a Likert scale from 1 (not true) to 5 (definitely true). The total score is the sum of responses and ranges from 7 to 35; higher scores indicate higher organizational priority.
Organizational Priority Measure Score | Month 22
  7-item assessment of organizational priority (adapted from Klein, et al.) administered to staff and rated on a Likert scale from 1 (not true) to 5 (definitely true). The total score is the sum of responses and ranges from 7 to 35; higher scores indicate higher organizational priority.
Organizational Priority Measure Score | Month 29
  7-item assessment of organizational priority (adapted from Klein, et al.) administered to staff and rated on a Likert scale from 1 (not true) to 5 (definitely true). The total score is the sum of responses and ranges from 7 to 35; higher scores indicate higher organizational priority.
Sustainment based on Fidelity Checklist Score | Month 15
  Sustainment of the overdose prevention practices will be measured using fidelity checklist score results. Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.
Sustainment based on Fidelity Checklist Score | Month 22
  Sustainment of the overdose prevention practices will be measured using fidelity checklist score results. Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.
Sustainment based on Fidelity Checklist Score | Month 29
  Sustainment of the overdose prevention practices will be measured using fidelity checklist score results. Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.
Sustainment based on Fidelity Checklist Score | Month 36
  Sustainment of the overdose prevention practices will be measured using fidelity checklist score results. Buildings will receive a fidelity checklist score of 0 (not implemented), 1 (partial implementation), or 2 (full implementation) for each overdose prevention practice. The primary outcome is total summed score, with higher scores indicating greater fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Doran, MD, MHS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified staff and tenant questionnaire data will be shared beginning 3 months and ending 5 years following article publication with qualified researchers who have a research question appropriate to the data and of potential benefit to permanent supportive housing tenants. Deidentified data will only be provided in aggregate after completion of a data use agreement (DUA). Requests should be directed to Kelly.Doran@nyulangone.org. All requests for such data will be presented to the study's Advisory Board for approval. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Qualified researchers who have a research question appropriate to the data and of potential benefit to permanent supportive housing tenants will be granted access to the data. Requests should be directed to Kelly.Doran@nyulangone.org. Deidentified data will only be provided in aggregate after completion of a data use agreement (DUA). All requests for such data will be presented to the study's Advisory Board for approval.

REFERENCES:
- [Derived] Gaeta Gazzola M, Torsiglieri A, Blaufarb S, Velez L, Hernandez P, O'Grady MA, Shelley D, Frank D, Cleland CM, Doran KM. Understanding overdose risk and response in permanent supportive housing: results of focus groups with tenants, staff, and leaders. Addict Sci Clin Pract. 2025 Nov 28;20(1):91. doi: 10.1186/s13722-025-00616-4. PMID 41316389
- [Derived] Doran KM, Torsiglieri A, Blaufarb S, Hernandez P, Melnick E, Velez L, Cleland CM, Neighbors C, O'Grady MA, Shelley D. The POP (Permanent Supportive Housing Overdose Prevention) Study: protocol for a hybrid type 3 stepped-wedge cluster randomized controlled trial. Implement Sci. 2023 Jun 7;18(1):21. doi: 10.1186/s13012-023-01278-z. PMID 37287026